CLINICAL TRIAL: NCT07329374
Title: Additional Effects of Ladder Drills and Jump Training on Agility, Core Stability and Balance of Taekwondo Players
Brief Title: Additional Effects of Ladder Drills and Jump Training in Taekwondo Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0482
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Sports Physical Therapy
Keywords: Ladder drills; Jump training; Taekwondo players

STUDY DESIGN:
Intervention Model Description: Randomized control design
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Intervention Group (Ladder Drills + Jump Training) The intervention plan consists of two main parts: Ladder Training and Jump Training, each lasting 20 minutes.
  Interventions: Other: Ladder drills; Other: Jump training
- Group B (Experimental): Control Group (Conventional Training) The control group plan will include 20 minutes of dynamic stretching and 20 minutes of aerobic training.
  Interventions: Other: Jump training

INTERVENTIONS:
Other: Ladder drills — The intervention plan consists ladder drills lasting 20 minutes.
  Arms: Group A
Other: Jump training — The intervention plan consists jump training lasting 20 minutes.

SUMMARY:
A Randomized controlled trial will be conducted with sample size of 40 players divided into two groups of 20, 20 players in each. Players will undergo 18 training sessions in six weeks, and each week has three training sessions. Each session, including a 10-minute warm-up and a 10-minute cool down, with 60 minutes in duration. The training will start with low intensity for the first two weeks, then progress to moderate intensity for the next two weeks, and finally reach high intensity, to the individual's ability and physical endurance.

DETAILED DESCRIPTION:
Taekwondo is a dynamic martial art that requires skill in speed, strength, flexibility, and coordination. It includes a variety of powerful techniques, such as kicks, punches, and defensive moves. For athletes to perform at their best and reduce the risk of injury, it is essential to develop flexibility, balance, and core strength. However, traditional Taekwondo training often emphasizes agility, instead of core stability and balance. The most basic drill involves jumping with one foot into each box of the ladder in motion forward and then the other foot in a quick manner. Jump training, especially plyometric training, is concerned with training the body to produce explosive force and speed, essential qualities in a taekwondo performer. To address this issue, the current study aims to explore the added benefits of combining ladder drills and jump training into a regular Taekwondo training program. This is a single-blinded, randomized controlled trial and will involve male Taekwondo athletes aged 18 to 25. Participants will be randomly assigned into two groups: Group A will receive standard Taekwondo training with ladder and jump drills, while Group B will focus on standard Taekwondo training only. This will be a 6-week training program consisting of a total of 18 sessions held 3 times a week. Each 60-minute session will include a 10-minute warm-up, 40 minutes of ladder drills and jump training, and a 10-minute cool-down phase. Data will be collected from athletes affiliated with the Pakistan Sports Board Lahore, focusing on three key variables: agility, core strength, and balance. These variables will be measured using standardized tests: the T-Test for agility, the Plank Test for core stability, and the Star Excursion Balance Test for balance. Assessments will be conducted before and after the training program to find changes in these physical characteristics. The results of this study will aim to assist coaches and trainers in enhancing Taekwondo performance while also focusing on injury prevention.

ELIGIBILITY:
Inclusion Criteria:

* Male Players
* Age 18-25 years
* Body mass index (BMI) between 20 and 30 kg/m2
* Participants with 1 year experience in Taekwondo

Exclusion Criteria:

* Players with any neurological disease that impairs balance or coordinated movement
* Participants will be involved in weight loss during the period of this study
* Current Musculoskeletal Injury
* Using any performance-enhancing drugs or supplements
* History of Lower Limb Injury or Surgery in the Past Year

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
T-Test for Agility | 6 weeks
  The T-Test takes 1-2 minutes per trial, and therefore 5-6 minutes for 2-3 trials. A typical arrangement of cones has 5m with the top of the Τ letter and 2.5m between them horizontally, while they are 9 to 12 inches high generally. Runners race ahead, make side-to-side movements to the left and right, then run backward to the starting line; the best agility scores are the shortest.
Core Stability Test | 6 weeks
  The Core Stability Test may take anywhere between 1 and 3 minutes per trial. Superior core stability is demonstrated in exercising athletes who undertake as long as possible for the forearm plank position.
Star Excursion Balance Test (SEBT) | 6 weeks
  The SEBT will measure dynamic balance by 2 to 3 minutes for each trial. Athletes stand on one leg and reach as far as possible in eight directions: forward, backward, inward, outward, forward-inward, forward-outward, backward-inward, and backward-outward.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Usman, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board coaching center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zemkova E, Zapletalova L. The Role of Neuromuscular Control of Postural and Core Stability in Functional Movement and Athlete Performance. Front Physiol. 2022 Feb 24;13:796097. doi: 10.3389/fphys.2022.796097. eCollection 2022. PMID 35283763
- [Background] Huang Z, Dai J, Chen L, Yang L, Gong M, Li D, Sun J. Effects of Progressive and Velocity-Based Autoregulatory Resistance Training on Lower-Limb Movement Ability in Taekwondo Athletes. Sports Health. 2025 May-Jun;17(3):545-555. doi: 10.1177/19417381241262024. Epub 2024 Aug 7. PMID 39109891
- [Background] Choi DS, Jung EN, Park MH. Comparison of balance ability and physical fitness according to the growth period in taekwondo players. J Exerc Rehabil. 2021 Oct 26;17(5):354-361. doi: 10.12965/jer.2142502.251. eCollection 2021 Oct. PMID 34805025
- [Background] Norjali Wazir MRW, Van Hiel M, Mostaert M, Deconinck FJA, Pion J, Lenoir M. Identification of elite performance characteristics in a small sample of taekwondo athletes. PLoS One. 2019 May 31;14(5):e0217358. doi: 10.1371/journal.pone.0217358. eCollection 2019. PMID 31150424
- [Background] Gabriel EH, Powden CJ, Hoch MC. Comparison of the Y-Balance Test and Star Excursion Balance Test: Utilization of a Discrete Event Simulation. J Sport Rehabil. 2020 Apr 23;30(2):214-219. doi: 10.1123/jsr.2019-0425. PMID 32325427
- [Background] Plesa J, Ujakovic F, Ribic A, Bishop C, Sarabon N, Kozinc Z. Effectiveness of an Individualized Training Based on Dynamic Strength Index on Sprinting, Jumping and Change of Direction Performance in Basketball Players: A Randomized Controlled Trial. J Sports Sci Med. 2024 Sep 1;23(1):504-514. doi: 10.52082/jssm.2024.504. eCollection 2024 Sep. PMID 39228784